CLINICAL TRIAL: NCT02574000
Title: Observational Study to Investigate Proportion of Patients With Hemiplegic Shoulder Pain Within 72 Hours Post-stroke and at Follow-up 8-10 Weeks Later.
Brief Title: Observational Study of Hemiplegic Shoulder Pain After Recent Stroke
Acronym: SPARS
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 15.0216
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Shoulder Pain; Hemiplegia; Stroke
MeSH Terms: conditions — Shoulder Pain; Hemiplegia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group baseline and follow-up: Single group of adult stroke patients assessed using ShoulderQ shoulder pain questionnaire and Clinical shoulder examination at two time-points:
  Baseline: within 72 hours post-stroke Follow-up: at 8-10 weeks post-stroke
  Interventions: Other: ShoulderQ which is a shoulder pain questionnaire; Other: Clinical shoulder examination

INTERVENTIONS:
Other: ShoulderQ which is a shoulder pain questionnaire — Questions regarding shoulder pain at rest, during movement and at night with visual analogue scales. Factors affecting shoulder pain.
Other: Clinical shoulder examination — Shoulder-Hand-Score (measuring pain, oedema, passive range of movement), muscle strength (using Oxford scale and National Institute of Health Stroke Scale (NIHSS) upper limbe motor and shoulder joint palpation (recording subluxation and soft-tissue pain).

SUMMARY:
This is an observational study to address the following questions.

1. How many people develop stroke-shoulder pain within 3 days of stroke?
2. How many people have stroke shoulder pain at 8-10 weeks after stroke?
3. Does having stroke-shoulder pain within 3 days of stroke predict the likelihood of having stroke-shoulder pain at 8-10 weeks?
4. What are the best bedside examination tests to identify stroke-shoulder pain?

DETAILED DESCRIPTION:
Patients will be assessed very early after stroke (within 72 hours) and followed up 8-10 weeks later. Findings will enable planning of fully-powered randomised controlled trials of both, pain-prevention strategies and treatment.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of haemorrhagic or ischaemic stroke

Exclusion Criteria:

* Transient Ischaemic attack,
* Neurological symptoms due to causes other than acute stroke,
* Unconscious,
* Severe behavioural disturbance,
* Severe agitation,
* Severe dementia,
* For palliation,
* Totally unable to communicate using any method - written, verbal, pictures, gesture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults within 72 hours of stroke
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline severity of hemiplegic shoulder pain at 8-10 weeks | within 72 hours and 8-10 weeks
  Questionnaire including visual analogue scales
Change from baseline Shoulder-Hand-Score at 8-10 weeks | within 72 hours and 8-10 weeks
  Measurement of pain, oedema, passive range of shoulder abduction and passive range of shoulder external rotation
Change from baseline NIH Stroke Score Upper limb (Motor Arm) at 8-10 weeks | within 72 hours and 8-10 weeks
  Muscle Strength
Change from baseline presence/absence of pain on palpation at 8-10 weeks | within 72 hours and 8-10 weeks
  Palpation of shoulder joint line and surrounding soft tissues
Change from baseline presence/absence of inferior glenohumeral subluxation at 8-10 weeks | within 72 hours and 8-10 weeks
  Palpable gap in sub-acromial region with arm dependent

CONTACTS AND LOCATIONS:
Overall Officials: Martine Nadler, PhD, Principal Investigator — St George's, University of London
Locations (1):
- St George's Hospital, Tooting, London, Greater London, United Kingdom

REFERENCES:
- [Background] Blennerhassett JM, Gyngell K, Crean R. Reduced active control and passive range at the shoulder increase risk of shoulder pain during inpatient rehabilitation post-stroke: an observational study. J Physiother. 2010;56(3):195-9. doi: 10.1016/s1836-9553(10)70025-4. PMID 20795926
- [Background] Gamble GE, Barberan E, Laasch HU, Bowsher D, Tyrrell PJ, Jones AK. Poststroke shoulder pain: a prospective study of the association and risk factors in 152 patients from a consecutive cohort of 205 patients presenting with stroke. Eur J Pain. 2002;6(6):467-74. doi: 10.1016/s1090-3801(02)00055-1. PMID 12413435
- [Background] Lindgren I, Jonsson AC, Norrving B, Lindgren A. Shoulder pain after stroke: a prospective population-based study. Stroke. 2007 Feb;38(2):343-8. doi: 10.1161/01.STR.0000254598.16739.4e. Epub 2006 Dec 21. PMID 17185637
- [Background] Ratnasabapathy Y, Broad J, Baskett J, Pledger M, Marshall J, Bonita R. Shoulder pain in people with a stroke: a population-based study. Clin Rehabil. 2003 May;17(3):304-11. doi: 10.1191/0269215503cr612oa. PMID 12735538
- [Derived] Nadler M, Pauls M, Cluckie G, Moynihan B, Pereira AC. Shoulder pain after recent stroke (SPARS): hemiplegic shoulder pain incidence within 72hours post-stroke and 8-10 week follow-up (NCT 02574000). Physiotherapy. 2020 Jun;107:142-149. doi: 10.1016/j.physio.2019.08.003. Epub 2019 Aug 9. PMID 32026814